CLINICAL TRIAL: NCT05269147
Title: Lidocaine Versus Bupivacaine for Sphenopalatine Ganglion Block in Patients Undergoing Endoscopic Septoplasty:A Comparative Study
Brief Title: Lidocaine Versus Bupivacaine for Sphenopalatine Ganglion Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huda Fahmy Mahmoud, PhD (Other)
Responsible Party: Sponsor-Investigator, Huda Fahmy Mahmoud, PhD, Assistant professor of Anaesthesia and Intensive Care department, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 506/1/21
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Septum; Deviation, Congenital
MeSH Terms: interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Intervention Model Description: To determine the efficacy of lidocaine versus bupivacaine for sphenopalatine ganglion block in patients undergoing endoscopic septoplasty.
  Postoperative Pain-free duration (minutes) will be recorded from the time of extubation to the first postoperative analgesic request when VAS ≥ 4 is the primary outcome.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SBGB with normal saline (Placebo Comparator): patients will receive standardized general anesthesia + SBGB with normal saline.
  Interventions: Procedure: Sphenopalatine Ganglion Block (SPGB)
- SBGB with lidocaine 2% (Active Comparator): patients will receive standardized general anesthesia + SBGB with lidocaine 2%
  Interventions: Procedure: Sphenopalatine Ganglion Block (SPGB)
- SBGB with bupivacaine 0.5% (Active Comparator): patients will receive standardized general anesthesia+ SBGB with bupivacaine 0.5%
  Interventions: Procedure: Sphenopalatine Ganglion Block (SPGB)

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block (SPGB) — The SPGB will be done after the patient is generally anesthetized and will be performed by the operating surgeon using a transnasal endoscopic approach through the posterior and over the middle turbinate tail in the pterygopalatine fossa.
  The patient will be placed in the supine position with head extension. The prepared solution (4 ccs 2% lidocaine or 0.5% bupivacaine or normal saline and 1 cc 8 mg dexamethasone) will be given (2,5 cc) to each side of the nose.
  The surgery was started 10 minutes after the application of SPBG to allow sufficient time for the block to develop.

SUMMARY:
The endoscopic septoplasty technique is one of the most frequently performed operations by otolaryngologists throughout the world. It is suggested that 86% of patients who undergo an endoscopic septoplasty would experience pain, and 75% of them suffer moderate to extreme levels of pain. Appropriate management of post-operative pain is a critical component of nasal surgery as it reduces perioperative morbidity, complications, hospital stay, and costs.

The sphenopalatine ganglion (SPG) is located in the cranial section of the autonomous nervous system; it is connected with the brain stem and the central nervous system (CNS) and bears unique characteristics favorable for the treatment of many painful syndromes involving the face and head. Sphenopalatine ganglion block (SPGB), along with general anesthesia (GA), is one of the regional anesthetic techniques used to reduce the need for systemic analgesia and provides relative hypotension with controlled heart rate that may lead to a better surgical field for endoscopic surgery. In addition, SPGB appears to shorten hospital stays and reduce narcotic requirements in the recovery area. SPGB with bupivacaine delivered repetitively appears to decreased postoperative pain and more satisfaction with the surgery for patients. Also, Bupivacaine usage in nasal surgery provides better analgesia at least in the first 8 hours period and does not cause more bleeding. On the other hand, SPGB with lidocaine was found to decrease the need for additional analgesics in the postoperative period, increase patient satisfaction, decrease the length of hospital stay, and as a consequence, reduce the rate of secondary infections. However, no previous studies have demonstrated the superiority of one drug over the other when performing an intranasal SPG block.

Aim of the work: To determine the efficacy of lidocaine versus bupivacaine for sphenopalatine ganglion block in patients undergoing endoscopic septoplasty.

DETAILED DESCRIPTION:
Methods:

Eligible patients will be evaluated by:

Preoperative:

Explanation of visual analog scale will be done to patients (the VAS consists of a straight, vertical 10-cm line; the bottom point represented "no pain" = (0 cm) and the top "the worst pain you could ever have" = (10 cm).

Randomization:

All patients fitting the inclusion criteria will be randomly allocated using computer-generated numbers into one of three groups. Labeled slips will be put in serially numbered opaque and sealed envelopes. They will be opened when an eligible patient will be enrolled by an independent worker, not worked in the study.

Group A (20 patients): patients will receive standardized general anesthesia + SBGB with normal saline.

Group B (20 patients): patients will receive standardized general anesthesia + SBGB with lidocaine 2% Group C (20 patients): patients will receive standardized general anesthesia+ SBGB with bupivacaine 0.5%

All patients will not receive anything per oral for at least 6 hours before a procedure. On arrival at the operation theatre, standard monitoring will be connected. Mean blood pressures (MBP), heart rate (HR) will be measured before the block (0 min.) and then every 10 minutes after the block till recovery time.

The patients will be received standardized GA protocol as follows:

1. Induction with propofol (1-2 mg/kg body weight),
2. Atracurium as a muscle relaxant (1 mg/kg body weight),
3. Isoflurane as a volatile anesthetic agent in 50% O2 and air, and
4. Analgesia with fentanyl (1 microgram/kg body weight). The total doses of fentanyl that were used during the operation will be recorded.

The patient will be evaluated intraoperatively and postoperatively for :

The Scoring criteria for an intraoperative surgical field using Fromme ordinal scale:

0 No bleeding

1. Slight bleeding but no suctioning of blood required
2. Slight bleeding with occasional suctioning required; surgical field not threatened
3. Slight bleeding with frequent suctioning required; bleeding threatens surgical field a few seconds after suction is removed
4. Moderate bleeding with frequent suctioning required; bleeding threatens the surgical field directly after suction is removed
5. Severe bleeding with constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery not possible

Postoperative Post-operative pain will be questioned by an anesthesiologist with a Visual Analog Scale (VAS) (0 = no pain, 10 = most severe pain) at the 30th minute(t1), 1st hour(t2), 4th hour (t3), 12th hour (t4) and 24th hours (t5) and analgesia was managed according to the VAS scores. If the VAS score is ≥ 4, the patient will be given rescue analgesia in the form of intravenously Pethidine 50mg.

The data on Postoperative nausea and vomiting will be collected by direct questioning by the anesthesiologist at the same time as pain score assessment. If there is 1 min between the episodes of vomiting, each one will be considered a separate episode. Every episode of vomiting will be scored as 1 point and the total score will be calculated after 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. The patients planned to perform endoscopic septoplasty
2. American Society of Anesthesiologists class I and II

Exclusion Criteria:

1. patients that will be received additional surgery with endoscopic septoplasty
2. patients under the age of 18
3. Patients have systemic or bleeding disorders
4. patients who disincline to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain-free duration (minutes) | 24 hours
  this time will be recorded from the time of extubation to the first postoperative analgesic request when VAS ≥ 4

SECONDARY OUTCOMES:
Postoperative Visual Analog Pain Score | 24 hours
  10 p0ints scale with 0 = no pain, 10 = most severe pain
Surgical field assessment from incision to closure | 3 hours
  assessment will done will performed using the Fromme ordinal scale, in which the surgeon grades the operating field from 0 (no bleeding) to 5 (severe bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: huda F fahmy, Principal Investigator — Aswan University
Locations (1):
- Huda Fahmy, Aswān, Egypt